CLINICAL TRIAL: NCT06073457
Title: Creation of Side-to-Side Compression Anastomosis Using the GT Metabolic Solutions Magnet System, GJ Biofragmentable to Achieve Gastro-Ileal or Gastro-Jejunal Diversion in Adults With Obesity
Brief Title: Magnetic Gastro-Ileal or Gastro-Jejunal Diversion Study ("MGI/MGJ Study")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GT Metabolic Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTM-003
Record Dates: First submitted 2023-07-17; First posted 2023-10-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A 2-stage, open-label, multicenter study enrolling up to 35 subjects at 6 study centers, as follows:
  * Stage 1: First-in-human (FIH) and proof-of-concept with up to 5 subjects; and
  * Stage 2: Feasibility with up to 30 subjects There will be a pause after completing enrollment in Stage 1 to allow completion of Day 30 and evaluation of safety by the independent Data Safety Monitoring Committee (DSMB). The DSMB will confirm whether the study can advance to Stage 2. All subjects in Stage 1 and 2 will be followed for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MagGJ System (Experimental): GT Metabolic Solutions Magnet System, GJ Biofragmentable ("MagGJ System")
  Interventions: Device: MagGJ System

INTERVENTIONS:
Device: MagGJ System — Anastomoses achieved by magnetic compression.

SUMMARY:
The purpose of this clinical research study is to evaluate the feasibility of the GT Metabolic Solutions Magnet System, GJ Biofragmentable ("MagGJ System") for creation of a side-to-side anastomosis for gastro-ileal or gastro-jejunal diversion in obese adults.

DETAILED DESCRIPTION:
The purpose of this clinical research study is to evaluate the feasibility of the GT Metabolic Solutions Magnet System, GJ Biofragmentable ("MagGJ System") for creation of a side-to-side anastomosis for gastro-ileal or gastro-jejunal diversion in obese adults. This partial diversion of intestinal contents from the stomach to the ileum or jejunum is intended to facilitate weight management/loss in obese adults and improve metabolic outcomes in obese adults with type 2 diabetes mellitus ("T2DM"). Side-by-side anastomoses are currently created by sutures, staples, and anastomotic compression devices. A predicate procedure is the single anastomosis sleeve ileal (SASI) bypass procedure that includes a gastro-ileostomy at the distal antrum of the stomach. Additionally, the one anastomosis gastric bypass (OAGB) or single anastomosis gastric bypass (SAGB) performed in two stages may also be considered a predicate procedure where an anastomosis between the jejunum and anterior lesser curvature of the stomach is performed, followed by a second stage gastric pouch stapling more than 12 months later (non-study procedure).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, inclusive, at the time of informed consent
* BMI 30-50 kg/m2, inclusive with either (A) Type 2 Diabetes Mellitus (T2DM), defined as HbA1c ≥ 6.5%, or (B) Weight regain following previous sleeve gastrectomy (>12 months) and indicated for a gastro-ileal diversion; OR
* BMI 35-50 kg/m2, inclusive without previous sleeve gastrectomy, and where (A) Gastro-jejunal diversion is indicated for the first stage, of a 2-stage, one anastomosis gastric bypass (OAGB), or (B) Single anastomosis gastric bypass (SAGB), with the second stage gastric pouch stapling performed >12 months after the gastro-ileal diversion, and not part of the investigational study
* Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for the duration of the study
* If a child-bearing female, subject must commit to not becoming pregnant and agree to use contraception for the duration of the study
* Willing and able to comply with protocol requirements

Exclusion Criteria:

* Type 1 diabetes
* Use of injectable insulin
* Uncontrolled T2DM
* Plan to perform a sleeve gastrectomy and/or hiatal hernia repair and/or cholecystectomy with the investigational study gastro-ileal anastomosis procedure
* Uncontrolled hypertension, dyslipidemia or sleep apnea
* Prior intestinal, colonic or duodenal surgery, other than bariatric
* Prior surgery, trauma, prostheses, disease or genetic expression which prevent or contra-indicate the procedure, including scarring and abnormal anatomy.
* Refractory gastro-esophageal reflux disease (GERD)
* Barrett's disease
* Helicobacter pylori positive and/or active ulcer disease
* Large hiatal hernia
* Inflammatory bowel or colonic diverticulitis disease
* Any anomaly precluding orogastric access by gastroscope and catheters, and manipulation techniques.
* Implantable pacemaker or defibrillator
* Psychiatric disorder, except well-controlled depression with medication for > 6 months
* History of substance abuse
* Woman who is either pregnant or breast feeding
* Woman of childbearing potential who does not agree to use an effective method of contraception.
* Any comorbidity or current status of subject's physiological fitness that in the surgeon's or anesthesiologist's opinion represents safety concerns that make the subject medically unfit for the procedure, including any significant congenital or acquired anomalies of the GI tract at or distal to the placement of the magnets.
* Unhealed ulcers, bleeding lesions, tumor, or any other lesion at target magnet deployment site
* Expected MR imaging within a two-month window following the study procedure
* Any anomaly preventing/contraindicating endoscopic or laparoscopic access and procedures
* Underwent a surgery/intervention within the 30 days proceeding the study procedure
* Any scheduled surgical or interventional procedure planned within 30 days post-study procedure
* Any stroke/TIA within 6 months prior to informed consent
* Requires chronic anticoagulation therapy (except aspirin)
* Active infections requiring antibiotic therapy, unless resolved before undergoing the study procedure
* Unable to comply with the follow-up schedule and assessments
* Recent tobacco or nicotine product cessation; cessation ≤ 3 months prior to informed consent
* Known allergies to the device components or contrast media
* Limited life expectancy due to terminal disease
* Currently participating in another clinical research study with an investigational drug or medical device
* A positive COVID-19 test prior to the study procedure, where indicated by local COVID-19 protocols for procedure/surgical clearance
* Any condition that, in the investigator's opinion, may preclude completion of follow-up assessments through Day 360 (e.g., a medical condition that may increase the risk associated with study participation or may interfere with interpretation of study results, inability to adhere to the visit schedule, or poor compliance with treatment regimen)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Magnet Placement | 1 Day
  MagGJ System placement ≥ 90% alignment of magnets
Natural Magnet Passage | 30 Days
  Passage of magnets without surgical re-intervention
Anastomosis Patency | Day 30
  Confirmed radiologically or fluoroscopically

CONTACTS AND LOCATIONS:
Locations (4):
- Westmount Surgical Center, Westmount, Quebec, Canada
- Clinica MEDS La Dehesa SpA, Santiago, Chile
- Hospital Lusiadas Amadora, Amadora, Portugal
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No